CLINICAL TRIAL: NCT01849523
Title: Web-based Tailored Information and Support for Patients With a Neuroendocrine Tumor: a Randomized Pilot Study (Pilot WIN-study).
Brief Title: Web-based Tailored Information and Support for Patients With a Neuroendocrine Tumor: a Randomized Pilot Study
Acronym: WIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pilot WIN-2013; NL43834.042.13 (Other: ABR number CCMO)
Record Dates: First submitted 2013-05-03; First posted 2013-05-08 (Estimated); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Distress; Quality of Life; Neuroendocrine Tumor
Keywords: Neuroendocrine tumor; Website; Information; Psychosocial support
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Web-based information and support (Experimental): Web-based tailored information and support
  Interventions: Behavioral: Web-based information and support
- Standard care (No Intervention): Standard care

INTERVENTIONS:
Behavioral: Web-based information and support
  Arms: Web-based information and support

SUMMARY:
Background Physical as well as psychosocial complaints are frequently present in patients with a neuroendocrine tumor (NET). Adequate information is seen as an essential aspect of supportive care. The aim of the current study is to test the effectiveness of a web-based tailored information and support system targeting patients' information and care needs. Key features of this system are self-screening of physical and psychosocial problems, tailored education on reported problems and self-referral to professional health care.

Objective To detect whether a web-based tailored information and support system improves patients' perception and satisfaction of received information. The investigators hypothesize that after having received web-based tailored information and support patients feel more informed and are more satisfied with the received information than when receiving standard care.

Study design The present study is a randomized prospective longitudinal experimental multicenter pilot study. In this study, we want to examine the effect sizes on the perception and satisfaction by the patient of received information (primary objective) and secondary objectives after having used web-based tailored information and support. Eligible are newly diagnosed NET-patients (N=40) (diagnosed less than 3 months ago). Patients will be asked to fill out questionnaires at baseline and after 12 weeks, on socio-demographic features (only at baseline), internet use (only at baseline), health care use, patients' perception and satisfaction of received information, distress, quality of life and empowerment (only after 12 weeks).

Study population Patients diagnosed with a NET (any type of NET, any phase of disease) who are under treatment at the Department of Medical Oncology in the University Medical Center Groningen or Hospital Medisch Spectrum; twenty will be invited to participate in the study.

Intervention During 12 subsequent weeks, a personalized website (with a surname/password) will become available to patients in the experimental group beside the usual standard care. Key features of the website are self-screening, tailored patient education and self-referral. Self-screening will be performed by an online version of the Dutch Distress thermometer (DT) and Problem List (PL). Patients will receive automated feedback on their DT score immediately after test completion together with information regarding problems reported on the PL, options for (self)-help and possibilities for referral to professional care. Contact information will also be available to discuss questions, problems and/or referral needs. Patients may also request a telephone call.

Main study endpoint The primary endpoint is to detect an improvement in patients' perception and satisfaction of received information after having received web-based tailored information and support.

ELIGIBILITY:
Inclusion Criteria:

* Adult NET patients (aged ≥ 18 years of age) with any tumor site and disease stage.
* Ability to comprehend Dutch (both reading and writing).
* Informed consent provided.

Exclusion Criteria:

* Estimated life expectancy less than 3 months.
* Patients with a second primary tumor for which active follow-up or treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-10; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
detect an improvement in perception and satisfaction of the received information | 14 weeks. This is the period a patient can use the website, thereafter a end-of study questionnaire will be filled out
  The primary objective is to detect an improvement in perception and satisfaction of the received information by NET-patients after having used the online tailored information and support system. We hypothesize that patients perceive to have received more information and are more satisfied with the received information after having used the web-based tailored information and support system.

SECONDARY OUTCOMES:
Distress level after receiving information | 14 weeks. This is the period a patient can use the website, thereafter a end-of study questionnaire will be filled out
  To test whether patients experience less distress after having received web-based tailored information and support.
Quality of life | 14 weeks. This is the period a patient can use the website, thereafter a end-of study questionnaire will be filled out
  To test whether patients experience a higher quality of life after receiving web-based tailored information and support.
Empowerment enhancement | 14 weeks. This is the period a patient can use the website, thereafter a end-of study questionnaire will be filled out
  To examine whether a web-based tailored information and support system enhances empowerment within the meaning of being better informed, feeling more confident in the relationship with their physician, improved acceptance of the illness, feeling more confident about the treatment and increased optimism and control over the future.

CONTACTS AND LOCATIONS:
Overall Officials: A.M.E. Walenkamp, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (2):
- Netherlands (2):
  - Medical Spectrum Twente, Enschede
  - University Medical Center Groningen, Groningen

REFERENCES:
- [Derived] Bouma G, de Hosson LD, van Woerkom CE, van Essen H, de Bock GH, Admiraal JM, Reyners AKL, Walenkamp AME. Web-based information and support for patients with a newly diagnosed neuroendocrine tumor: a feasibility study. Support Care Cancer. 2017 Jul;25(7):2075-2083. doi: 10.1007/s00520-017-3598-7. Epub 2017 Feb 9. PMID 28185086